CLINICAL TRIAL: NCT00735631
Title: Evaluation of the Accuracy, Safety and Robustness of a Single-input-single-output (SISO) Model-based Predictive Closed-loop System to Guide Patient-individualized ICU Sedation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/489
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Coronary Artery Disease
Keywords: Patients entering the post-operative cardiac intensive care unit following coronary artery reconstruction surgery.
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The single-input-single-output (SISO) model-based predictive closed-loop system will be used to guide patient-individualized ICU sedation with propofol
  Interventions: Device: SISO model-based predictive closed-loop system

INTERVENTIONS:
Device: SISO model-based predictive closed-loop system — The single-input-single-output (SISO) model-based predictive closed-loop system will be used to guide patient-individualized ICU sedation with propofol

SUMMARY:
The aim of this study is to investigate the accuracy, safety and robustness of a single-input-single output (SISO) model-based predictive closed-loop system to guide patient-individualized ICU sedation.

ELIGIBILITY:
Inclusion Criteria:

* patients in the immediate post-operative phase after an coronary artery reconstruction surgery.
* age >= 18 years
* informed consent obtained before the surgery

Exclusion Criteria:

* severe renal failure defined by the RIFLE Classification levels Risk, Failure and End-stage Kidney Failure
* severe hepatic failure defined by a bilirubin level of >= 3 mg/dl and/or a prothrombin level of < 50% before the surgery
* low ejection fraction defined as < 40%
* age < 18 years
* postoperative bleeding so that a new surgery is necessary
* history of cardiovascular accident (CVA)
* history of COPD
* age > 75 years
* postoperative cardiac index < 2.2 for more than 2 hours
* SvO2 < 60% for more than 2 hours
* hypotension with a MAP < 60 mmHg for more than 2 hours
* sedation agents other than remifentanyl and propofol including also Catapressan, Risperdal, Etumine
* Remifentanyl dose exceeding 0.5 µg/kg/min.
* absence of informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The propofol and remifentanil dose needed to keep the BIS within the target range | During sedation

SECONDARY OUTCOMES:
The hemodynamic stability of the patient, being defined as: - mean arterial blood pressure between 65 and 85 - heart rate around 80 beats'/min - diuresis 0.5 - 1 ml/kg/hour - normal pH - normal cardiac index as defined by a CI > 2.2 - Sv02 > 60 % | During sedation

CONTACTS AND LOCATIONS:
Overall Officials: Michel Struys, MD, PhD, Principal Investigator — University Hospital, Ghent; Annick De Wolf, MD, Principal Investigator — University Hospital, Ghent; Johan Decruyenaere, MD, PhD, Principal Investigator — UIniversity Hospital Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Neckebroek M, Ionescu CM, van Amsterdam K, De Smet T, De Baets P, Decruyenaere J, De Keyser R, Struys MMRF. A comparison of propofol-to-BIS post-operative intensive care sedation by means of target controlled infusion, Bayesian-based and predictive control methods: an observational, open-label pilot study. J Clin Monit Comput. 2019 Aug;33(4):675-686. doi: 10.1007/s10877-018-0208-2. Epub 2018 Oct 11. PMID 30311073
- See also: Website of the University Hospital Ghent — http://www.uzgent.be